CLINICAL TRIAL: NCT07289009
Title: Adaptation and Implementation of the InterRAI-HC System Used in Home Health Care Services in Turkish
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, İkbal Oğuz Karaalp, Registered Nurse, PhD Candidate, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HU-HF-IOK-01
Record Dates: First submitted 2025-11-26; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Home Health Care
Keywords: Home Health Care; Older Adults; Nursing Care; Quality of Life

STUDY DESIGN:
Intervention Model Description: The study is designed methodological research. The first stage is the validity-reliability stage. In the second stage, a randomized controlled trial will be conducted to measure the effectiveness of the adapted scale. The intervention group will receive care using the adapted scale, while the control group will receive standard care.
Masking Description: Participants included in the study will be assigned to intervention and control groups using a stratified randomization method based on the home health care units to which their caregivers belong. To ensure homogeneity between groups, "care unit and participant age" will be taken into account. Participants will first be stratified by age and care unit. Which group will be included in the Turkish validity and reliability study of the InterRAI-HC application (intervention) or the comparison of the InterRAI scale with standard forms (control) will be determined by lottery before assignment. Group "A" represents the InterRAI-HC application group, and group "B" represents the control group. To prevent selection bias, randomization will be performed using a sequence of random integers generated by a bio-statistician independent of the study using a computer. Participants will then be assigned to the intervention (n=18) and control (n=18) groups using simple randomization. Neither participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care-Centered Group (Experimental): Scale-focused care will be provided to this group. The care process will be maintained using care plans developed by the researcher based on literature information, including NANDA diagnoses, NIC interventions, and NOC outcomes.
  Interventions: Behavioral: Care supports
- Control Group (No Intervention): This group will receive standard nursing care.

INTERVENTIONS:
Behavioral: Care supports — The intervention of the study involves providing nursing care to the elderly individual and caregivers using care plans designed by the researcher, utilizing a validated scale. The adapted scale provides a comprehensive geriatric assessment. Emerging issues will be evaluated using NANDA diagnoses and NIC interventions/NOC outcomes. Individuals in the intervention group will be followed up for 6 months with these care plans. No interventions other than the services provided under ESH will be performed on individuals in the control group. The adapted questionnaire and specified scales will be administered simultaneously at the initial interview (0 months) and at 6 months for individuals in this group.
  Other Names: individual-centered nursing care
  Arms: Care-Centered Group

SUMMARY:
This study was designed with a methodological approach. The first phase of the study consists of establishing the validity and reliability of the "International Resident Assessment Instrument-Home Care (InterRAI-HC)" application in Turkish. The second phase of the study involves comparing the standard forms used in Home Health Services units with the adapted InterRAI scale. The study population will consist of caregivers of individuals aged 65 and over who apply to the home health services unit of a healthcare institution in Kars province. The interRAI-HC questionnaire, SF-12 scale, and nursing care plans will be used to collect data. The aim of the study is to develop a comprehensive geriatric assessment tool for use in home health services.

DETAILED DESCRIPTION:
Advances in healthcare technology, the focus of planned policies on disease prevention, and the expansion of healthcare services to wider areas have resulted in longer life expectancy, bringing with it other problems that need to be addressed. Therefore, the goal of "healthy aging," defined as a process of aging that enables individuals to maintain their physical fitness, achieve mental and physical balance, become self-sufficient, contribute to the welfare of society with their existing abilities, and remain independent into old age, has been included in the planned policies. In line with this goal, the WHO published the "European Healthy Aging Strategy and Action Plan 2012-2020," and Turkey also published the "Turkey Healthy Aging Action Plan and Implementation Program 2021-2026" . According to 2023 data from the Turkish Statistical Institute (TÜİK), the countries with the highest elderly populations are Monaco, Japan, and Italy, respectively. According to 2023 data from the Turkish Statistical Institute, the elderly population rate in Turkey is 10.2%. The same report states that an elderly population ratio above 10% indicates population aging. According to the TUİK 2023 report, there are 8 million 722 thousand elderly people in Turkey, and 1 million 669 thousand of them live alone. Considering both the burden of disease and current employment conditions in the literature, and based on projections that the elderly population ratio will be 16.3% in 2040, the elderly are seen as the community most in need of home care . The purpose of home health services is to protect the individual's health and aim to improve their quality of life, to ensure that impaired health is regained to the maximum extent possible, and to be in constant communication with the elderly individual and their family. In this context, home health services are characterized as services that reduce or delay the length of stay in institutions. Sources in the literature report that the development of home health services within the scope of elderly care services has led to a decrease in hospital admissions and frequent repeat hospitalizations. The most important feature of home health services is that they aim to achieve these goals in the individual's home environment while involving family members in care to the maximum extent possible. International literature indicates that individuals prefer to have their care needs met at home. Similarly, according to the 2023 TÜİK report, 31.6% of elderly people in Turkey stated that they wanted to live while receiving home care services. In light of these data, it is evident that the elderly population is more eager for care services in the home environment and that the burden of care will increase for home care services.

Research has shown that due to factors such as rising healthcare costs, limited bed capacity in healthcare facilities, and, as noted in the literature, individuals' freedom of choice, providing care services in individuals' homes, where they feel safer and more comfortable, rather than in healthcare facilities, has become a new generation goal . Looking at examples of home healthcare services around the world, India, which has the largest population after China, established a "National Policy for the Elderly" in 2011 and developed the concept of "aging in place." Under this policy, the concept of home-based care services was adopted through state and private institutions. Germany, one of the European countries with the largest elderly population, is among the countries that advocate that care services should be provided primarily in the home environment during the aging process. For this reason, the interRAI-International Resident Assessment Instrument, a comprehensive tool for home care service planning, is used. This test assesses the individual's mobility, self-sufficiency, cognitive status, and communication skills, and plans the care services they will need. In Finland, where the elderly population constitutes 23% of the total population, the KATI (Smart Aging and Home Care) program aims to support healthy aging at home. This program provides early diagnosis services using artificial intelligence applications developed with technology, preventing diseases and ensuring the development of a long-term care approach without the need for institutional care .In our country, the "Regulation on the Provision of Home Health Services by the Ministry of Health and Affiliated Institutions," published in the Official Gazette (No. 29280) on February 27, 2015, provides for the organization of home health services under hospitals, municipalities, oral and dental health hospitals, and community health centers. The care services provided include hospital-based practices such as dressing changes, simple examinations, and some intravenous and intramuscular procedures, while early diagnosis services or psychosocial support practices are provided to a limited extent.

In planning for healthy aging, another issue as important as establishing the units where the service will be provided is ensuring the quality and continuity of care. Therefore, it is necessary to conduct a comprehensive geriatric assessment for each individual receiving this service, to accurately record and store this information, to ensure information sharing within or between institutions through a multidisciplinary work plan, to plan interventions related to existing multiple diseases, to be prepared for sudden changes that may occur with aging, and to develop action plans for crisis management.In this context, the use of standardized data for data collection and planning in home health care has become even more important in providing high-quality care. Considering the requirements for quality care, interRAI, which provides a series of standardized comprehensive assessments covering multiple domains and aims to improve the care process for every individual in the community, is actively used by both researchers and practitioners in 35 countries. A retrospective cohort study conducted in Ontario, Canada, in 2022 measured the impact of the interRAI-HC application on emergency visits. The results of this research reported that comprehensive interRAI-HC assessments can identify potential emergencies in individuals in advance and reduce emergency visits. A study conducted in New Zealand indicated that the interRAI system can create a common language among healthcare professionals and enable a multidisciplinary team approach in elective surgical situations and palliative care admissions. A 2023 study in Ireland indicated that interRAI assessment tools are effective in identifying the needs of family caregivers. The interRAI system, whose effectiveness has been proven in many countries, has five different areas that collect and measure data on specific topics. These are stated as home health, long-term care, mental health, care for individuals with developmental and intellectual disabilities, and child and adolescent mental health. Looking at the literature on home health among these areas; In a study conducted. Visits made using the interRAI-Home Care (interRAI-HC) application, which they customized for use in home care services between 2001 and 2014, the characteristics of the elderly individuals visited, and the patient-oriented results of the system were shared. According to this study, over a 10-year period, patients with declining cognitive and functional abilities received more visits than other patients. The same study also showed that the identification of increasing frailty led to the planning of new health policies and extended the period during which the care needs of elderly individuals could be met in a home environment. In a systematic review conducted by Salahudeen and Nishtala in 2019, it was stated that the interRAI-HC application is effective in determining admission indications and assessing caregiver burden, in addition to comprehensive geriatric assessment, and that it can play an effective role in making key decisions regarding the care process. In our country, the scales used for healthy aging have been designed or integrated by independent researchers and their effectiveness has been proven. However, when looking at current health practices, there is no measurement tool that provides a comprehensive geriatric assessment officially used by healthcare providers. In this context, there is a need for a system that helps improve the quality and continuity of healthcare by conducting comprehensive geriatric assessments in our country, storing this data, sharing it with relevant individuals or organizations, and planning interventions.

Hypotheses and Objectives Underlying the Thesis Proposal The aim of this study is to develop and implement a version of the InterRAI-HC application, which is part of the InterRAI system used in many areas in 35 countries, that is suitable for use in Turkey.

1. Research Questions Is the InterRAI-HC scale a reliable tool for ensuring continuity of care for individuals receiving home care services in Turkish society? Is the InterRAI-HC scale a valid tool for ensuring continuity of care for individuals receiving home care services in Turkish society?
2. Research Design The research was planned in a methodological design.
3. Data Collection Tools The following tools were used to collect data: the InterRAI-HC questionnaire, the Short Form (SF)-12, and the Standard Forms used in HHS (Home Health Services) will be used.
4. Implementation Study Sample and The Validity and Reliability Study of the InterRAI-HC Scale This includes the steps for adapting the scale to Turkish and Turkish culture. The adaptation process includes language validity, construct validity, content validity, and reliability stages.

   The study population consists of 700 elderly individuals who meet the inclusion criteria. The literature reports that 5-10 times the number of items is sufficient for validity and reliability analysis. InterRAI-HC consists of 45 scale items. A 10% loss rate was added to the number, aiming to reach 250 individuals. At this stage, InterRAI questionnaire owners were consulted, and advice was sought on the adequacy of this number. At this stage, data will be collected from individuals receiving health services themselves or from informal caregivers by formal caregivers.
5. Sample and Implementation of the Intervention Study To determine whether there is a difference between two independent groups, the Independent Samples T-Test will be used under the assumption of normality. Accordingly, the sample size of the study was determined by considering the mean and standard deviations of the 12-month results of the Pain sub-dimension in the "Nurse Care Coordination in Community-Based Long-Term Care" study. The sample size of the study was calculated using the G*Power 3.1.9.2 software package. Accordingly, the minimum sample size required for 80% power at a 0.05 significance level and 0.976 effect size was determined to be 36 (18 elderly individuals per group).

   5.1. Intervention Group The literature indicates that the InterRAI assessment should be repeated at three-month intervals. Therefore, it was deemed appropriate to conduct three face-to-face interviews: the first interview (month 0), the third month, and the sixth month. These interviews will be planned as home visits on days scheduled with Home Health Services, and assessments will be provided. The care process of the individuals will be carried out simultaneously by HHS personnel and researchers.

   5.2.Control Group No intervention other than the services provided under HHS will be made to the individuals in the control group. The developed questionnaire and defined scales will be applied to individuals in this group simultaneously at the first meeting (0 months) and at 6 months.
6. Randomization and Prevention of Bias Participants included in the study will be assigned to the intervention and control groups using a stratified randomization method based on the home health care units to which their caregivers belong. "Care unit and participant age" will be taken into account to ensure homogeneity between groups. Participants will first be stratified by age and care unit. Which group will be included in the Turkish validity and reliability study of the InterRAI-HC application (intervention) or the comparison of the InterRAI scale with standard forms (control) will be determined by lottery before assignment. Group "A" represented the InterRAI-HC application group, and group "B" represented the control group. To prevent selection bias, randomization will be performed using a sequence of random integers generated by a bio-statistician independent of the study using a computer. Participants will then be assigned to the intervention (n=18) and control (n=18) groups using simple randomization. Neither participant nor investigator blinding will be applied in the study.

ELIGIBILITY:
Inclusion criteria;

* Being registered with ESYS (Home Health Care Management System),
* Volunteering to participate in the study
* Having a caregiver

Exclusion criteria:

• Not knowing Turkish

Withdrawal criteria from the study:

* Refusing two or more scheduled visits,
* Withdrawing at the individual's own request,
* Providing incomplete or incorrect responses.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
SF-12 | 6 months
  The SF-36 Scale consists of 12 selected questions from the SF-36 Questionnaire. In 1992, the Rand Corporation developed and released the SF-36 Health Survey. Koçyiğit and colleagues established its validity and reliability in Turkish. The SF-12 consists of eight subscales. Scores ranging from 0 to 100 can be obtained from the scale. Higher scores indicate a higher quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Harakani State Hospital, Kars, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No